CLINICAL TRIAL: NCT05777538
Title: Effects of Foot Exercises With and Without Hydrotherapy on Pedal Edema & Lower Extremity Function in Antenatal Women
Brief Title: Effects of Foot Exercises and Hydrotherapy on Pedal Edema & Lower Extremity Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0511
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: foot; exercises; hydrotherapy; pedal; edema lower extremity; antenatal; women
MeSH Terms: conditions — Motor Activity | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot exercise with hydrotherapy (Experimental): Hydrotherapy will be performed by immersing the women's foot in a container filled with 3 liters water with a temperature of 30-32°C. The water level must cover the women's feet up to ankle. During the immersion the therapist will ask the women to perform exercise with legs being fully supported, then alternatively stretch and flex the ankle for 30 times. which will be followed by circling each foot at ankle in clock wise and anticlock wise direction, 30 times each. The duration of water immersion session will be (30 min) for 5 consecutive days
  Interventions: Other: hydrotherapy; Other: foot exercises
- Foot exercise (Active Comparator): The therapist will ask the women to perform exercise with legs being fully supported, then alternatively stretch and flex the ankle for 30 times. which will be followed by circling each foot at ankle in clock wise and anticlock wise direction, 30 times each
  Interventions: Other: foot exercises

INTERVENTIONS:
Other: hydrotherapy — Hydrotherapy will be performed by immersing the women's foot in a container filled with 3 liters water with a temperature of 30-32°C. The water level must cover the women's feet up to ankle. During the immersion the therapist will ask the women to perform exercise with legs being fully supported, then alternatively stretch and flex the ankle for 30 times. which will be followed by circling each foot at ankle in clock wise and anticlock wise direction, 30 times each. The duration of water immersion session will be (30 min) for 5 consecutive days.
  Arms: Foot exercise with hydrotherapy
Other: foot exercises — The therapist will ask the women to perform exercise with legs being fully supported, then alternatively stretch and flex the ankle for 30 times. which will be followed by circling each foot at ankle in clock wise and anticlock wise direction, 30 times each.

SUMMARY:
To determine the Effects of foot exercises with and without hydrotherapy on pedal Edema & lower extremity function in antenatal women.

ELIGIBILITY:
Inclusion Criteria:

* Normal singleton pregnancy
* Gestational age 30-40 weeks
* Pitting edema in feet

Exclusion Criteria:

* presence of any under lying disease e.g.

  * Diabetes,
  * Hypertension,
  * High risk pregnancy
  * Any wound or skin lesion

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant female
Enrollment: 44 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Figure of 8 Method | 8th week
  The figure of 8 method uses landmarks on the foot and ankle to measure the circumference of ankle in centimeters.
  1. the point midway over the anterior ankle between the tibialis anterior tendon and lateral malleolus,
  2. the navicular tuberosity,
  3. the base of the fifth metatarsal, and
  4. the inferior tip of the medial malleolus
Lower Extremity Functional Scale | 8th week
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used to evaluate the functional status of lower limb

CONTACTS AND LOCATIONS:
Overall Officials: Hina gul, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Sajida Khalil Hospital Gujrat, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] .MACWAN KR, Savaliya PK. Effectiveness of Foot Exercise and Epsom Salt Water on Reduction of Foot Oedema among Antenatal Mothers. Journal of Clinical & Diagnostic Research. 2021;15
- [Background] Talbot L, Maclennan K. Physiology of pregnancy. Anaesthesia & Intensive Care Medicine. 2016;17(7):341-5
- [Background] Patola A, Tridiyawati F. The Effectiveness of Soaking the Feet in Salt Water to Reduce the Degree of Edema in Pregnant Women Trimester III. Jurnal Keperawatan Komprehensif (Comprehensive Nursing Journal). 2022;8
- [Background] Ahmed AH, Ismail NIAA, Hassan NMM. Effect of effleurage massage versus water immersion with exercise on physiological foot edema among primigravidae. Egypt J Health Care. 2021;12(2):56-345